CLINICAL TRIAL: NCT04718714
Title: Effects of Dexmedetomidine vs Propofol on Inflammatory Response and Intra-abdominal Pressure in Patients With Intra-abdominal Sepsis; a Randomized Clinical Trial
Brief Title: Effects of Dexmedetomidine vs Propofol in Patients With Intra-abdominal Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ibraheem Abdelmageed, assistant lecturer at anaesthesia and ICU department faculty of medicine assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00008718
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Septic Peritonitis
MeSH Terms: interventions — Midazolam; Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- midazolam (Active Comparator): postoperative ventilation and sedation with continuous intravenous infusion of midazolam only for 24 hours
  Interventions: Drug: Midazolam
- propofol (Active Comparator): postoperative ventilation and sedation with continuous intravenous infusion of propofol only for 24 hours
  Interventions: Drug: Propofol
- dexmedetomidine (Experimental): postoperative ventilation and sedation with continuous intravenous infusion of dexmedetomidine only for 24 hours
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — loading dose intravenous infusion of 0.2 mg/kg over 10 minutes followed by a maintenance dose of 0.02 -0.2 mg /kg/hr. over 24 hours.
  Arms: midazolam
Drug: Propofol — loading dose intravenous infusion of one mg/kg over 15 minutes followed by a maintenance dose of 20-80 microgram/kg/min. over 24 hours.
  Arms: propofol
Drug: Dexmedetomidine — loading dose of dexmedetomidine of one µg/kg over 10 minutes followed by maintenance dose of 0.2 -1.5 µg/kg/hr. over 24 hours.
  Arms: dexmedetomidine

SUMMARY:
Sepsis is defined as systemic response to infection ,and it is a main problem in ICU and despite advance in supportive care, the mortality rate in patients with severe sepsis continues to exceed 30% [Bone RC 1993].The effects of bacterial invasion of body tissues result from combined actions of enzymes and toxins produced by micro-organisms themselves and by a network of proinflammatory mediators and cytokines as tumour necrosis factor α and interleukin 6 which are overexpressed after various noxious insults[P.Delong et al. 2006],[ Yealy et al. 2014].

the patients who are subjected to abdominal surgery in order to treat the cause surgically,and many of these surgical procedures are lengthy and are at risk for either pre-operatively or post-operatively with steady increase in intra-abdominal pressure(IAP) [Malbrain ML et al. 2007] Intra-abdominal hypertension (IAH) is defined as IAP equal to or greater than 12 mmHg whereas abdominal compartment syndrome (ACS) is defined as IAP greater than 20 mmHg, abdominal perfusing pressure (APP) is used to predict prognosis of both IAH and ACS [Malbrain ML et al. 2006].

The choice for using a sedative agent in ICU for mechanically ventilated patients post-operatively is therefore a crucial one as these patients are under hyperstress state and often require drugs for sedation and analgesia[ Chanques G et al. 2006].

Analgesics and sedation agents have clearly been shown to alter cellular function and other mediators of immune system with wide range of immune modulation ,ranging from immunosuppressive effects to significant anti-inflammatory effects during endotoxaemia[ Taniguchi et al. 2004] Also sedation and /or analgesia have the potential to reduce IAP through improvement of abdominal wall compliance.

Although propofol and dexmedetomidine are used for sedation in ICU there are limited data on their effects on inflammatory responses and IAP in septic patients.

In clinical practice, septic patients treated with dexmedetomidine have shorter time on the ventilator as compared with those treated with lorazepam, a benzodiazepine and this beneficial effect of dexmedetomidine is more pronounced in septic patients than in nonseptic patients. This outcome may be partly the result of dexmedetomidine induced reduction in pulmonary inflammatory mediators and lung tissue damage.[ M. Ueki et al. 2014] Midazolam is known to inhibit certain aspects of the immune function. It was suggested that benzodiazepines bind to specific receptors on macrophages and inhibit their capacity to produce IL-1, IL-6, and TNFα.

Propofol, nowadays, has become a preferred sedative in ICU because it offers advantages over benzodiazepines in terms of lack of accumulation, quick onset, easy adjustment, and fast recovery after discontinuation. [ Jacobi J et al. 2002]

DETAILED DESCRIPTION:
After surgery patients will be transferred to the ICU and will be randomly allocated by use of sealed envelopes ;into one of three groups 20 patients each.

All ICU measurements will be recorded by an observer

The following data will be collected:

* Patients' demographic and clinical data including age, sex, weight ,operative procedure time and type and patient's SOFA score.
* Mean arterial pressure, heart rate (HR), central venous pressure (CVP), and temperature will be continuously monitored . Urine output will be measured hourly and fluid balance will be calculated every 12 hours. All measurements will be obtained at the start of the study (baseline), then at the 24th and 48th hours.
* Lactate, platelets, leukocytes, bilirubin, alanine aminotransferase, and creatinine will be determined at the same times TNF-α, IL-1β, and IL-6 levels will be obtained at baseline, and at the 24th and 48 th hours.
* Intraabdominal pressure and abdominal perfusion pressure will be measured at baseline (15 min before start of the study) and at the 24th and 48th hours per the study protocol.
* Behavioral pain scale, ramsay sedation score and post operative analgesics requirements as a rescue analgesia.
* Duration of mechanical ventilation and length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* patients aged18 years old or more and had the criteria of intraabdominal sepsis as evident by quick sofa score of 2 or more and have done intraabdominal surgical procedures

Exclusion Criteria:

* children pregnant women Patients who receive neuromascular blockers during the first 48 hours of ICU admission known allergy or contraindication to propofol ,dexemedetomidine or midazolam known or suspected brain death

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-23 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
interleukin 1 plasma concentration | 48 hours
  interleukin 1 plasma concentration will be measured three times, at admission ,24 hours after admission and 48 hours after admission
interleukin 6 plasma concentration | 48 hours
  interleukin 6 plasma concentration will be measured three times ,at admission ,24 hours after admission and 48 hours after admission
intraabdominal pressure per mmHg | 48 hours
  intraabdominal pressure will be measured three times ,at admission ,24 hours after admission and 48 hours after admission

SECONDARY OUTCOMES:
difference of mean time of ventilator free days | 28 days
  difference of mean time of ventilator free days between the three arms

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No